CLINICAL TRIAL: NCT02549352
Title: Efficacy and Safety of LEO 43204 in Field Treatment of Actinic Keratosis on Balding Scalp Including 12-month Follow-up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0084-1196
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2018-12

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 43204 gel (Experimental): Treatment once daily for 3 days
  Interventions: Drug: LEO43204 gel
- Vehicle gel (Placebo Comparator): Treatment once daily for 3 days
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: LEO43204 gel
  Other Names: Ingenol Disoxate
  Arms: LEO 43204 gel
Drug: Vehicle gel
  Arms: Vehicle gel

SUMMARY:
The objective of the trial is to compare the short term efficacy of LEO 43204 gel with vehicle gel in AK on the balding scalp when applied topically once daily for 3 consecutive days as field treatment

ELIGIBILITY:
Inclusion Criteria:

* Subjects with 5 to 20 clinically typical, visible and discrete AKs within a treatment area of sun-damaged skin on the full balding scalp (the balding part of the scalp should be greater than 25 cm2 (4 in2) and up to approximately 250 cm2 (40 In2)
* Subjects with minimum 3 clinically typical, visible and discrete AKs within a tracking area of 50 cm2 (8 In2). The tracking area must be within the treatment area

Exclusion Criteria:

* Location of the treatment area (balding scalp) within 5 cm of an incompletely healed wound or within 5 cm of a suspected BCC or SCC
* Treatment with ingenol mebutate gel in the treatment area within the last 12 months
* Lesions in the treatment area that have: atypical clinical appearance (e.g. hyperthrophic, hyperkeratotic or cutaneous horns) and /or, recalcitrant disease (e.g. did not respond to cryotherapy on two previous occasions)
* History or evidence of skin conditions other than the trial indication that would interfere with the evaluation of the trial medication (e.g. eczema, unstable psoriasis, xeroderma pigmentosum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09-22 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf-Markus Szeimies, Prof. Dr.med, Principal Investigator — Klinik für Dermatologie & Allergologie Klinikum Vest GmbH
Locations (1):
- Klinik für Dermatologie & Allergologie Klinikum Vest GmbH, Recklinghausen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 391 participants were enrolled, 80 were screening failures, and 311 participants were randomized. Only 310 of the randomized participants were treated with investigational medicinal product (IMP), the number of participants treated is reflected as the number of participants started in the first period.
Groups:
- LEO 43204 0.037% Gel: Treatment once daily with LEO 43204 0.037% gel for 3 consecutive days applied on the scalp.
- Vehicle Gel: Treatment once daily with vehicle gel for 3 consecutive days applied on the scalp.
Period: 3-day Treatment and 8-week Follow-up
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Started | 209 | 102
Treated | 209 | 101 (1 participant was included in 0.037% in the safety analysis set as they received both IMPs in error)
Completed | 207 | 96
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Other | 0 | 2
Period: 12-month Follow-up
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Started | 207 | 93
Completed | 199 | 81
Not Completed | 8 | 12
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 3 | 2
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel | Total
Number analyzed (Participants) | 209 | 101 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (9.0) | 71.0 (9.3) | 70.1 (9.1)
Age, Customized [Count of Participants; unit: Participants]
  Age group: 18-64 years | 60 | 17 | 77
  Age group: 65-84 years | 139 | 75 | 214
  Age group: >=85 years | 10 | 9 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 209 | 101 | 310
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 45 | 25 | 70
  Italy | 23 | 12 | 35
  United States | 141 | 64 | 205

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Clearance of Actinic Keratosis (AK)
Description: The number of clinically visible actinic keratosis lesions (AKs) identified in the treatment area was recorded at Day 1 (baseline), Weeks 4, and 8.
  Complete clearance was defined as no clinically visible AKs in the treatment area.
  The table shows the percentage of mean number of participants across imputations with complete clearance at Week 8.
Time Frame: At Week 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Number analyzed (Participants) | 209 | 101
percentage of participants | 22.0 [16.4 to 27.7] | 3.0 [-0.3 to 6.3]
Statistical Analysis 1: Comparison: LEO 43204 0.037% Gel vs Vehicle Gel; Test type: Superiority; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 7.83, 95% CI 2-sided [2.58 to 23.71] — Mantel-Haenszel estimate (0.037% relative to vehicle), adjusted for pooled sites

2. Secondary Outcome: Percentage of Participants With Partial Clearance
Description: The number of clinically visible Actinic keratosis lesions (AKs) identified in the treatment area was recorded at Day 1, Weeks 4, and Week 8.
  Partial clearance was defined as at least 75% reduction from baseline in the number of clinically visible AKs in the treatment area.
  The table shows the percentage of mean number of participants across imputations with partial clearance at Week 8.
Time Frame: At Week 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Number analyzed (Participants) | 209 | 101
percentage of participants | 63.1 [56.5 to 69.7] | 11.0 [4.9 to 17.2]
Statistical Analysis 1: Comparison: LEO 43204 0.037% Gel vs Vehicle Gel; The p-values for secondary endpoints have been corrected by the Holm-Bonferroni method to account for multiplicity. The prespecified multiplicity adjustment by the Holm-Bonferroni method requires the ordering of the p-values for the secondary endpoints by size; Test type: Superiority; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 5.91, 95% CI 2-sided [3.32 to 10.51] — Mantel-Haenszel estimate (0.037% relative to vehicle), adjusted for pooled sites

3. Secondary Outcome: Percentage of Participants With Partial Clearance
Description: The number of clinically visible Actinic keratosis lesions (AKs) identified in the treatment area was recorded at Day 1, Weeks 4, and Week 8.
  Partial clearance was defined as at least 75% reduction from baseline in the number of clinically visible AKs in the treatment area.
  The table shows the percentage of mean number of participants across imputations with partial clearance at Week 4.
Time Frame: At Week 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Number analyzed (Participants) | 209 | 101
percentage of participants | 53.4 [46.5 to 60.3] | 7.1 [2.0 to 12.1]
Statistical Analysis 1: Comparison: LEO 43204 0.037% Gel vs Vehicle Gel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 7.59, 95% CI 2-sided [3.70 to 15.61] — Mantel-Haenszel estimate (0.037% relative to vehicle), adjusted for pooled sites

4. Secondary Outcome: Percent Reduction in AK Count in the Treatment Area Compared to Baseline
Description: The percent reduction at Week 8 from baseline was analysed using a negative binomial regression for the AK count at Week 8 with treatment group and pooled sites as factors and baseline count as offset variable (using multiple imputations to account for missing values). The table presents adjusted mean percent reduction at Week 8 from baseline.
Time Frame: At Week 8
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Number analyzed (Participants) | 209 | 101
percentage of change | 74.0 [70.6 to 77.1] | 13.7 [0.2 to 25.3]
Statistical Analysis 1: Comparison: LEO 43204 0.037% Gel vs Vehicle Gel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel — Negative binominal regression with treatment group and pooled site as factors and log baseline count as offset variable; Week 8 AK count ratio = 0.30, 95% CI 2-sided [0.25 to 0.36] — 0.037% relative to vehicle

ADVERSE EVENTS:
Time Frame: Treatment period including follow-up (from Day 1 to Week 8) and extended follow-up (from Week 8 up to Month 14)
Description: Adverse events presented in the table are investigator-reported terms. Adverse events of special interest within system organ class (SOC) Neoplasm benign, malignant and unspecified (incl cysts and polyps), were adjudicated by an Independent Adjudication Committee based on central biopsy review.
  For further details on the adjudication outcomes, see link to the full report in section "More information"
  Adverse events are reported with a >=2% frequency threshold for the active treatment group.
Groups:
- LEO 43204 0.037% Gel - Extended Follow-up: Treatment once daily with LEO 43204 0.037% gel for 3 consecutive days applied on the scalp.
- Vehicle Gel - Extended Follow-up: Treatment once daily with vehicle gel for 3 consecutive days applied on the scalp.
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel | LEO 43204 0.037% Gel - Extended Follow-up | Vehicle Gel - Extended Follow-up
Serious Adverse Events (participants affected / at risk) | 3/210 | 3/100 | 0/208 | 0/92
Other Adverse Events (participants affected / at risk) | 146/210 | 12/100 | 5/208 | 1/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 43204 0.037% Gel (N=210) | Vehicle Gel (N=100) | LEO 43204 0.037% Gel - Extended Follow-up (N=208) | Vehicle Gel - Extended Follow-up (N=92)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 43204 0.037% Gel (N=210) | Vehicle Gel (N=100) | LEO 43204 0.037% Gel - Extended Follow-up (N=208) | Vehicle Gel - Extended Follow-up (N=92)
Application site pain (General disorders) | 118 | 3 | 1 | 0
Application site pruritus (General disorders) | 68 | 8 | 1 | 0
Eyelid oedema (Eye disorders) | 9 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 9 | 0 | 0 | 0
Eye irritation (Eye disorders) | 5 | 0 | 0 | 0
Headache (Nervous system disorders) | 11 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 15 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.